CLINICAL TRIAL: NCT04728581
Title: Mirtazapine and Quetiapine as Treatment for Postoperative Sleep Disturbance After Fast-track Knee Replacement
Brief Title: Improving Sleep After TKA Using Mirtazapine and Quetiapine
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Anna Ziekenhuis, Geldrop, Netherlands (Other)
Responsible Party: Principal Investigator, Walter van der Weegen, PhD, St. Anna Ziekenhuis, Geldrop, Netherlands
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: W021-001
Record Dates: First submitted 2021-01-12; First posted 2021-01-28 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-06

CONDITIONS: Osteo Arthritis Knee; Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Mirtazapine; Quetiapine Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): use of placebo during first 2 weeks after TKA surgery
  Interventions: Drug: Placebo
- Low dose Mirtazapine (Experimental): Use of Mirtazapine 3.75mg before lights-out, allowed to increase medication to 7.5mg
  Interventions: Drug: Mirtazapine
- Low dose Quetiapine (Experimental): use of Quetiapine 3.125mg before lights-out, allowed to increase medication to 6.25mg
  Interventions: Drug: Quetiapine

INTERVENTIONS:
Drug: Mirtazapine — Use of 3.75mg mirtazapine before lights-out during first 2 weeks after TKA surgery. With insufficient effect on sleep, patients are allowed to increase medication to 7.5mg mirtazapine.
  Arms: Low dose Mirtazapine
Drug: Quetiapine — Use of 3.125mg quetiapine before lights-out during first 2 weeks after TKA surgery. With insufficient effect on sleep, patients are allowed to increase medication to 6.25mg mirtazapine.
  Arms: Low dose Quetiapine
Drug: Placebo — a gelatinous capsule without an active ingredient
  Arms: Placebo

SUMMARY:
Use of mirtazapine and quetiapine for improvement of sleep quality after TKA

DETAILED DESCRIPTION:
Background After knee replacement surgery there is a loss of quantity and quality of sleep. Loss of sleep is associated with increased pain perception. Subsequently, patients use more analgesic medication and it takes them longer to fully recover from surgery. Low doses of the tetracyclic antidepressant mirtazapine and the neuroleptic quetiapine are nowadays off-label prescribed for insomnia and improve length and quality of deep sleep phases. Quetiapine and mirtazapine could improve sleep after knee replacement surgery and improve patient recovery. This placebo-controlled, randomized, double-blind study investigates the effect of quetiapine and mirtazapine on functional recovery after total knee arthroplasty.

Methods This is a prospective, single center, double-blinded randomized controlled trial. 165 patients with knee osteoarthritis scheduled for total knee arthroplasty will be randomly allocated to a low-dose quetiapine (LDQ), a low-dose mirtazapine (LDM) group or a placebo group. Outcomes will be evaluated at baseline, 2, 4, 6 and 12 weeks after surgery. Functional outcome after total knee arthroplasty is measured using a patient related outcome measure through the Oxford Knee Score (OKS). In order to measure postoperative sleep quality, patients will be monitored using the Leeds Sleep evaluation questionnaire (LSEQ). Furthermore, pain is registered using a visual analogue scale (VAS), weekly opioid use is monitored, and general health status is reported through the EQ-5D. Analyses will be conducted on an intention-to-treat basis using logistic and linear mixed regression models. This trial complies with the SPIRIT guidelines for randomized controlled trials.

Discussion This study will provide clinicians with evidence whether quetiapine contributes to rehabilitation of patients undergoing fast-track knee replacement surgery.

ELIGIBILITY:
Inclusion Criteria:

* Indication for TKA

Exclusion Criteria:

* use of benzodiazepines
* use of anti-depressants
* use of oxycodone
* patients diagnosed with obstructive sleep apnea syndrome, severe respiratory insufficiency, or myasthenia
* a known hypersensitivity to mirtazapine, quetiapine and/or related to the gelatinous (placebo) capsule
* insufficient understanding of the Dutch language.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Oxford Knee Score (OKS) | 6 weeks after surgery
  Validated functional knee score after TKA, minimum score 12 (best outcome), maximum score 60 (worst outcome)

SECONDARY OUTCOMES:
Leeds Sleep Evaluation questionnaire (LSEQ) | 1 week before surgery; first day postoperative; 2; 4; 6; 12 weeks after surgery
  Validated sleep score in 3 dimensions of sleep
Visual Analogue Scale (VAS) for fatigue | 1 week before surgery; first day postoperative; 2; 4; 6; 12 weeks after surgery
  Visual analogue reporting of fatigue after sleep, indicated on a 0 (best outcome) to 100 (worst outcome) mm line
Visual Analogue Scale (VAS) for sleep quality | 1 week before surgery; first day postoperative; 2; 4; 6; 12 weeks after surgery
  Visual analogue reporting of quality sleep, indicated on a 0 (worst outcome) to 100 (best outcome) mm line
Visual Analogue Scale (VAS) for pain in rest | 1 week before surgery; first day postoperative; 2; 4; 6; 12 weeks after surgery
  Visual analogue reporting of knee pain while resting, indicated on a 0 (best outcome) to 100 (worst outcome) mm line
Visual Analogue Scale (VAS) for pain during activity | 1 week before surgery; first day postoperative; 2; 4; 6; 12 weeks after surgery
  Visual analogue reporting of knee pain during exercises, indicated on a 0 (best outcome) to 100 (worst outcome) mm line
EuroQol (EQ) 5D | 1 week before surgery; first day postoperative; 2; 4; 6; 12 weeks after surgery
  General well being score, full health represented by 11111 score (overall score for the Netherlands of 1,000), worst health represented by 55555 score (overal score for the Netherlands of -0,329)
Morphine use | 1 week before surgery; first day postoperative; 2; 4; 6; 12 weeks after surgery
  Total amount (mg) morphine use after surgery is documented
Oxford knee score | 1 week before surgery; first day postoperative; 2; 4; 12 weeks after surgery
  Validated functional knee score after TKA, minimum score 12 (best outcome), maximum score 60 (worst outcome)

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Knowledge Center for Orthopedic Surgery, St. Anna hospital, Geldrop
  - St. Anna hospital, Geldrop

IPD SHARING:
Plan to Share IPD: Yes
All data free accessible upon request
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: First year after publication
Access Criteria: After written request, and received permission